CLINICAL TRIAL: NCT07049549
Title: Evaluation of the Effectiveness of Adjunctive Injectable Platelet-Rich Fibrin Application to Root Surface Debridement in Phase 1 Treatment of Smoking Patients With Periodontitis
Brief Title: The Effectiveness of Root Planing and Injectable Platelet-Rich Fibrin in Smoking Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Tolga Sönmez, research assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-KAE-0072
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Periodontal Healing; Periodontitis; i-PRF
Keywords: i-prf; periodontitis; root planing; platelet-rich fibrin; periodontal debridement
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: A split-mouth design will be used. Each subject would receive both interventions in selected (randomized) quadrants.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Active Comparator): Subjects would receive full-mouth scaling and root planing (SRP). Following instrumentation, autologous injectable platelet-rich fibrin (i-PRF) will be prepared from venous blood and administered subgingivally to the test quadrants according to a split-mouth design.
  Interventions: Biological: Injectable PRF
- Control Group (Placebo Comparator): Subjects will be receive full-mouth scaling and root planing (SRP). Following instrumentation, placebo (sterile saline) is administered subgingivally to the control quadrants according to a split-mouth design.
  Interventions: Other: Plasebo (Sterile Saline)

INTERVENTIONS:
Biological: Injectable PRF — Autologous injectable platelet-rich fibrin (i-PRF) will be prepared from venous blood using low-speed centrifugation and administered subgingivally to the test quadrants following full-mouth scaling and root planing.
  Arms: Test Group
Other: Plasebo (Sterile Saline) — sterile saline solution will be administered subgingivally to the control quadrants following full-mouth scaling and root planing (SRP).
  Arms: Control Group

SUMMARY:
Periodontitis is a chronic, multifactorial inflammatory disease characterized by the progressive destruction of the tissues supporting the teeth, associated with dysbiotic plaque biofilms. The foundation of non-surgical periodontal treatment is the mechanical debridement of the tooth surfaces to reduce bacterial load. In this phase, dental calculus and bacterial deposits are removed, and root surfaces are smoothened. This helps eliminate the microorganisms responsible for inflammation. Following treatment, epithelial healing occurs in the form of long epithelial attachment, which re-forms within approximately one week. The reduction of inflammatory cells, tissue repair, and decreased gingival crevicular fluid flow lead to the resolution of clinical signs such as redness and swelling. A tissue recession of 1-2 mm is generally observed. The fibrils in the connective tissue are altered or lysed during the disease process, and their reorganization and healing may take several weeks.

The aim of this study is to evaluate the clinical effects (plaque index, gingival index, bleeding on probing, probing pocket depth, clinical attachment level) of injectable platelet-rich fibrin (I-PRF) in addition to non-surgical periodontal treatment in periodontitis patients with deep pockets and smoking habits.

In advanced cases, surgical treatments may be required. According to the study by Heitz-Mayfield and colleagues, surgical treatment in pockets deeper than 6 mm resulted in a 0.6 mm greater reduction in probing depth and 0.2 mm more clinical attachment gain compared to scaling and root planing alone. However, for pockets between 4-6 mm in depth, non-surgical treatment resulted in 0.4 mm more attachment gain compared to surgical procedures. In a systematic review by Labriola and colleagues, it was found that smokers had a lesser reduction in pocket depth. Furthermore, Scabbia and colleagues reported that smokers had significantly lower clinical improvements after surgical treatment. Smoking negatively affects healing, and factors such as exposed root surfaces and protected areas for residual plaque contribute to disease recurrence. Long-term studies have shown that smokers experience higher tooth loss.

The use of blood-derived products in wound healing started 40 years ago, with fibrin adhesives standing out. Fibrin is the activated form of fibrinogen, a plasma molecule, and is the final product of coagulation. Polymerized fibrin forms the initial scar matrix in the wound area, serving as a biological adhesive that aids in hemostasis.

One of the most commonly used blood-derived products in dentistry is platelet-rich fibrin (PRF). Developed by Choukroun in 2001, this second-generation product can be prepared without anticoagulants, thrombin, or gelling agents. It is a simple and cost-effective method. Injectable PRF (I-PRF) is obtained by altering the centrifugation speed and duration. Miron and colleagues demonstrated that low-speed I-PRF contains a higher number of regenerative cells and growth factors. A study by Kour and colleagues showed that I-PRF has antimicrobial effects against periodontal pathogens such as Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans.

In conclusion, I-PRF, prepared from the patient's own blood, may provide biological support to non-surgical periodontal treatment, positively influencing the healing process and reducing the need for surgical interventions. The aim of this study is to assess the clinical effects (plaque index, gingival index, bleeding on probing, pocket depth, clinical attachment level) of I-PRF in conjunction with non-surgical periodontal treatment in periodontitis patients with deep pockets and smoking habits.

A total of 25 volunteers will be included in the study. Inclusion criteria are: not pregnant, no use of antibiotics, anti-inflammatory drugs, or systemic corticosteroids, no periodontal treatment in the past 6 months, presence of at least 20 teeth, bleeding on probing in ≥30% of sites, and at least two non-adjacent teeth in each quadrant with probing depth ≥5 mm, clinical attachment loss ≥4 mm, and radiographic evidence of bone loss in the coronal third (horizontal and/or vertical). Informed consent will be obtained after explaining the study.

Eligible participants will undergo clinical periodontal evaluation including plaque index (Silness & Löe, 1964), gingival index (Löe & Silness, 1963), probing depth, clinical attachment loss, and bleeding on probing (Ainamo & Bay, 1975). At the second visit, full-mouth scaling and root planing will be performed. In the test sites, injectable platelet-rich fibrin (I-PRF), prepared by centrifugation at 700 rpm for 3 minutes, will be applied. Control sites will receive saline without antimicrobial or regenerative effects. Follow-ups for oral hygiene reinforcement will be scheduled at 1 week, 1 month, and 3 months. Clinical measurements will be repeated at 3 months.

DETAILED DESCRIPTION:
Periodontitis is a chronic, multifactorial inflammatory disease characterized by the progressive destruction of tooth-supporting tissues associated with dysbiotic plaque biofilms. The loss of periodontal support manifests clinically as attachment loss, alveolar bone loss, periodontal pocket formation, and gingival bleeding. Due to its high prevalence, potential to cause tooth loss, negative impact on chewing function and esthetics, and reduction in quality of life, periodontitis is considered a significant public health concern. The primary etiological factor of the disease is microbial plaque and its byproducts.

The goal of periodontal treatment is to halt disease progression by controlling the microbial etiology and associated risk factors and to restore lost periodontal structures, thus maintaining a functional and esthetically acceptable dentition. Various treatment modalities have been developed to reduce bacterial plaque on root surfaces. Conventional methods include mechanical plaque removal using hand instruments and ultrasonic devices, with scaling and root planing considered the gold standard in periodontal therapy.

Adjunctive use of local agents with root surface debridement has shown additional benefits. These agents help reduce bacterial contamination and promote healing. Local antimicrobial agents suppress subgingival microbiota and support the control of inflammation. Other materials, such as hyaluronic acid and statins, have also demonstrated beneficial clinical outcomes when used in conjunction with non-surgical periodontal therapy.

Smoking is a major risk factor both for the onset of periodontitis and for a reduced treatment response. Smokers tend to exhibit less favorable healing after non-surgical treatments and experience greater tooth loss over time. Additionally, smoking can result in exposed root surfaces and protected areas that facilitate plaque accumulation, contributing to disease recurrence.

Platelets have gained attention in regenerative therapies due to their ease of collection and their rich content of growth factors. Platelet-derived factors such as TGF-β1 exhibit both pro- and anti-inflammatory properties. Platelets become activated following endothelial injury and, through various adhesion molecules, initiate inflammatory responses and support tissue repair. They also play a key role in hemostasis and wound healing by stimulating fibroblast, endothelial, and progenitor cell activity through their released growth factors.

Platelet concentrates are classified into two generations: first-generation platelet-rich plasma (PRP) and second-generation platelet-rich fibrin (PRF). PRP preparation is complex, requiring additives and multiple centrifugation steps, and its clinical effect is limited by the rapid release of growth factors. PRF, in contrast, is a fully autologous product obtained by simple centrifugation of venous blood without additives. A variation known as injectable PRF (I-PRF), prepared at lower speeds and shorter durations, contains not only platelets and leukocytes but also stem and endothelial cells, thus being referred to as a "blood concentrate."

I-PRF has been shown to release higher levels of growth factors, enhance fibroblast migration, and increase the expression of collagen and regenerative cytokines. Additionally, I-PRF demonstrates stronger antimicrobial activity against periodontal pathogens compared to other platelet concentrates.

A total of 25 volunteers will be included in the study. Inclusion criteria are: not pregnant, no use of antibiotics, anti-inflammatory drugs, or systemic corticosteroids, no periodontal treatment in the past 6 months, presence of at least 20 teeth, bleeding on probing in ≥30% of sites, and at least two non-adjacent teeth in each quadrant with probing depth ≥5 mm, clinical attachment loss ≥4 mm, and radiographic evidence of bone loss in the coronal third (horizontal and/or vertical). Informed consent will be obtained after explaining the study.

Eligible participants will undergo clinical periodontal evaluation including plaque index (Silness & Löe, 1964), gingival index (Löe & Silness, 1963), probing depth, clinical attachment loss, and bleeding on probing (Ainamo & Bay, 1975). At the second visit, full-mouth scaling and root planing will be performed. In the test sites, injectable platelet-rich fibrin (I-PRF), prepared by centrifugation at 700 rpm for 3 minutes, will be applied. Control sites will receive saline without antimicrobial or regenerative effects. Follow-ups for oral hygiene reinforcement will be scheduled at 1 week, 1 month, and 3 months. Clinical measurements will be repeated at 3 months.

The aim of this study is to evaluate the clinical effects (plaque index, gingival index, bleeding on probing, probing pocket depth, and clinical attachment level) of adjunctive injectable platelet-rich fibrin application in non-surgical periodontal therapy in periodontitis patients with deep pockets who smoke.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years
* Having at least 20 natural teeth
* Presence of interproximal CAL and/or buccal or lingual CAL ≥3 mm accompanied by PPD >3 mm in at least two non-adjacent teeth
* Presence of periodontal pockets ≥4 mm in at least one site in each dental arch
* Smoking more than 10 cigarettes per day
* Absence of systemic diseases or ongoing medication use
* No antibiotic, anti-inflammatory, or systemic corticosteroid use within the last 6 months
* No periodontal treatment within the last 6 months
* Not pregnant, lactating, or menstruating

Exclusion Criteria:

* presence of systemic or oral diseases
* regular systemic medication use
* recent periodontal or pharmacological treatment history
* hormonal conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
The evaluation of changes in Probing Pocket Depth (PPD) | Baseline and 3 months
  Probing Pocket Depth (PPD) measurements are take at baseline (first session) and at the 3-month follow-up to assess clinical changes over time. Using a periodontal probe, the distance between the gingival margin and the base of the sulcus or periodontal pocket is measured at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatal/lingual, midpalatal/lingual, and distopalatal/lingual. Care is taken to keep the probe parallel to the long axis of the tooth and to apply minimal force during measurement. The values from the six sites are summed and divided by six to calculate the average PPD.
The evaluation of changes in Clinical Attachment Levels (CAL) | Baseline and 3 months
  CAL measurements are taken at baseline (first session) and at the 3-month follow-up to assess clinical changes over time. Using a periodontal probe, the distance between the enamel-cement junction and the base of the sulcus or periodontal pocket is measured at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatal/lingual, midpalatal/lingual, and distopalatal/lingual. The values from these six points are summed and divided by six to calculate the average clinical attachment level.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University, Faculty of Dentistry, Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No